CLINICAL TRIAL: NCT06287034
Title: The Role of the Free/Pedunculated Flap in Total Laryngectomy After (Chemo-)Radiotherapy Failure for Laryngeal Carcinoma: Impact on the Risk of Pharyngocutaneous Fistula (PCF)
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1833/23
Record Dates: First submitted 2024-01-12; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Larynx Carcinoma
Keywords: pharyngocutaneous fistula
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Salvage total laryngectomy STL primary suture: Patients in both groups will then undergo salvage total laryngectomy STL surgery with primary suturing.The primary suture can be performed according to the different techniques available at the discretion of the surgeon (vertical, horizontal or T-shaped closure, with continuous suture, according to Connell or with detached stitches)31. It would be preferable for all centers to use a homogeneous pharyngeal suture technique, such as the T-shaped with Connell suture.
  Interventions: Procedure: Primary suture
- Salvage total laryngectomy STL primary suture + onlay flap: Patients in both groups will then undergo salvage total laryngectomy STL surgery with primary suturing, but in the patients of the second group, in addition, the positioning of a free/pedunculated covering flap will also be carried out with the onlay technique. Reconstruction with the onlay technique can be performed using a pedicled pectoralis major myofascial flap or anterolateral thigh myofascial free flap at the surgeon's discretion (pharyngeal suture unchanged). The flap will be positioned with an onlay technique to reinforce the pharyngeal suture and in turn sutured to the prevertebral fascia or residual surrounding tissues.
  Interventions: Procedure: Primary suture

INTERVENTIONS:
Procedure: Primary suture — The primary suture can be performed according to the different techniques available at the discretion of the surgeon (vertical, horizontal or T-shaped closure, with continuous suture, according to Connell or with detached stitches)

SUMMARY:
Multicenter, prospective, randomized study aimed at evaluating the difference in risk of PCF after salvage laryngectomy in two groups of patients: one cohort treated with Total Laryngectomy (LT) with primary suture, a second group treated with LT and reinforcement by flap positioning with onlay technique (PMM, ALT)

DETAILED DESCRIPTION:
Patients, once eligibility has been verified, will then be randomized (1:1) to one of the following groups: Gruop 1: STL primary suture. Group 2: STL primary suture + onlay flap Patients in both groups will then undergo surgery STL with primary suture; in those of the second group, in addition, the positioning of a free/pedunculated covering flap will also be carried out with the onlay technique. 4 months after surgery, questionnaires will be administered to the patient for the subjective evaluation of the quality of life in relation to vocal rehabilitation obtained through voice prosthesis or esophageal voice (SECEL questionnaire) and swallowing rehabilitation (SOAL questionnaire). Demographic and preoperative data will be collected, data relating to pre-(chemo-)radiotherapy and pre-STL clinical staging, as well as the interval in days between the end of (chemo-)radiotherapy and surgery, perioperative data, type of eventual unilateral or bilateral laterocervical lymph node emptying, the type of pharyngotomy suture, the type of flap possibly used, the packaging of the tracheoesophageal fistula for positioning the voice prosthesis, the definitive histological examination.

The patient must undergo a radiological examination for loco-regional and distant staging before the STL (CT or MRI) and a biopsy demonstrating the recurrence/persistence of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of recurrence/persistence of squamous cell carcinoma of the larynx previously subjected to exclusive radiotherapy or concomitant chemo-radiotherapy treatment:

  1. pre (ChT-)RT staging: cT1/T2/T3 N0/N+;
  2. pre STL staging: rcT1/cT2/ Selected cT3 cT4a (extension to thyroid cartilage and/or prelaryngeal tissues) N0/N+ (clinically and radiologically).
* Indication for STL surgery (no pharyngeal mucosal resection);
* Functional total laryngectomies after radical (chemo-)radiotherapy treatment;
* Age > 18 years;
* Signature of informed consent and ability to complete in-office questionnaires.

Exclusion Criteria:

* STL extended to the pharynx and/or total pharyngeal laryngectomies;
* Extension of the tumor to the pharyngeal mucosa and/or massive extra-laryngeal extension;
* Previous open organ preservation surgery (OPHL).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from recurrence/persistence of laryngeal SCC following exclusive RT treatment or concomitant RT/ChT without extension to the pharynx (rcT1/T2/T3 selected rcT4a N0/N+) who will have to undergo STL and who will meet the following criteria. Patients undergoing extensive laryngectomies or with disease with even partial involvement of the pharyngeal mucosa (pyriform sinus, posterior wall of the pharynx) will not be included.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-03-21 (Estimated); Study Completion 2025-09-21 (Estimated)

PRIMARY OUTCOMES:
questionnaires for evaluation of the quality of life | 30 months
  Questionnaires will be administered to the patient for the subjective evaluation of the quality of life in relation to vocal rehabilitation obtained through voice prosthesis or esophageal voice (SECEL questionnaire).

SECONDARY OUTCOMES:
Identification of risk factors | 4 months
  Identification of risk factors related to the formation of pharyngocutaneous fistulas after salvage total laryngectomy
Evaluation of swallowing function | 4 months
  Evaluation of swallowing function assessed using the SOAL questionnaire
Evaluation of vocal rehabilitation | 4 months
  Evaluation of vocal rehabilitation using the SECEL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Raul Pellini, Doctor, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy